CLINICAL TRIAL: NCT07248007
Title: Effect of Platelet-Rich Plasma Injection on Wound Healing After Fistulotomy for Simple Anal Fistula Randomized Controlled Trial (RCT)
Acronym: PRPIWHAFSAFRCT
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Osama Ahmed, Demonstrator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RPRFISULOTOMY
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: Simple Anal Fistula
Keywords: anal fistula
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Intervention Model Description: comparison between 2 groups of patients with simple anal fistula one group use PRP with fistulotomy in treatment and the other group only do fistulotomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRP injection (Active Comparator): a group of patients with simple anal fistula that will be treated with PRP following fistulotomy
  Interventions: Procedure: PRP injection
- Non PRP group (No Intervention): the other group that will be treated with fistulotomy only without PRP

INTERVENTIONS:
Procedure: PRP injection — Injection of PRP after fistulotomy in simple low anal fistula
  Arms: PRP injection

SUMMARY:
Anal fistula is a common benign anorectal condition characterized by an abnormal tract between the anal canal and perianal skin, often resulting from cryptoglandular infection. Surgical fistulotomy remains the standard treatment for simple low anal fistulas, with success rates exceeding 90% .

However,wound healing following fistulotomy can be prolonged,ranging from 6-10 weeks,which affects patient comfort, quality of life, and return to normal activity (1,2).

After a fistulotomy, the tract is laid open, leaving behind a raw wound extending from the anal canal to the perianal skin.Traditionally,this wound is left open to heal by secondary intention(granulation and epithelialization).

In marsupialization, the cut wound edges (the mucosa and anoderm/skin) are sutured to the wound base.Thismakesthewoundshallowerandkeepsitopenfordrainage.Itpreventsadeepcavitythat would otherwise take longer to granulate and epithelialize.

Marsupialization of the wound edges has been introduced as a modification of standard fistulotomy to improve healing outcomes. Several randomized trials have shown that marsupialization accelerates wound healing (by 1-4 weeks) and preserves sphincter function better compared to leaving the wound open, without increasing recurrence or complications (3,4,5).

DETAILED DESCRIPTION:
Platelet-rich plasma(PRP) has been widely investigated and applied in several surgical fields because of its ability to promote tissue regeneration and accelerate healing. In orthopedic surgery, PRP has been used to enhance bone and tendon healing, particularly in the managementofchronictendinopathiesandfractures.Inplastic and reconstructive surgery,it has been applied to improve graft take, flap survival, and cosmetic outcomes in wound coverage.In maxillofacial and dental surgery, PRP has shown benefits in bone regeneration, implant integration, and periodontal healing. More recently, colorectal and general surgery have explored PRP for difficult-to-heal wounds, including anal fistula, where it has been demonstrated to shorten healing time and reduce recurrence rates

ELIGIBILITY:
Inclusion Criteria:

* Age18-65years. Both males and females. Clinical diagnosis of simple low anal fistula(confirmed by examination±imaging).

Simple fistula is defined as:

Fistula affecting less than one third of anal sphincter Fistula willnot affect sphincter function after surgery(no risk for fecal incontinence).

All types of low fistula which will not affect anal continence after surgery.

Exclusion Criteria:

* Complex or high anal fistulas:

( multiple tracts, suprasphincteric, extrasphincteric, or high transsphincteric tracts.) -Underlying diseases that impair healing: (Crohn's disease, ulcerative colitis, tuberculosis, HIV infection, anorectal malignancy)

* Hematological disorders: coagulopathy, thrombocytopenia, or platelet dysfunction.
* Systemic factors:

Uncontrolled diabetes mellitus. Immunosuppressive therapy (e.g., steroids, chemotherapy). Previous surgery for anal fistula (to avoid bias from scar tissue and recurrence)..

-Known allergy to any agents used in PRP preparation (rare, e.g., calcium chloride).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Operative time | intra operative
  messure the improvement of operative time between the PRP group and the non PRP group

SECONDARY OUTCOMES:
Post operative pain | 12 months
  messure the improvement of post operative pain between the 2 groups using the VIsual Analogue Scale (VAS) score